CLINICAL TRIAL: NCT06571006
Title: Effect of Music Therapy Applied During Lumbar Puncture on Infants' Pain Perception: Randomized Controlled Study
Brief Title: Effect of Music Therapy Applied During Lumbar Puncture on Infants' Pain Perception
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Erzurum Technical University (Other)
Responsible Party: Principal Investigator, Ayşe Metin, Assist. Prof., Erzurum Technical University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 227
Record Dates: First submitted 2024-08-19; First posted 2024-08-26 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: Infant ALL
Keywords: lumbar puncture; Infant; pain
MeSH Terms: conditions — Pain | interventions — Music Therapy

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experiment group (Experimental): The musical intervention will start 10 minutes before the lumbar puncture procedure begins and continue for another 20 minutes after the intervention. Babies will be kept away from noise during this study. W.A. It was decided to use the piece "Adagio" from the Violin Concerto No. 3 in G major, KV 216, composed by Mozart. The track will be played through two speakers on opposite sides, 30 cm away from the baby's ears, to optimize sound perception. High quality digital audio will be used to make babies listen. Music will be played at a level that can be heard in high noise pollution (i.e. the noise of incubator operation and the white noise of the recorder), but taking into account the permissible sound level recommended by the American Academy of Pediatrics, i.e. 65-70 dB.
  Interventions: Other: music
- control group (No Intervention): no intervention

INTERVENTIONS:
Other: music — The musical intervention will start 10 minutes before the lumbar puncture procedure begins and continue for another 20 minutes after the intervention. Babies will be kept away from noise during this study. W.A. It was decided to use the piece "Adagio" from the Violin Concerto No. 3 in G major, KV 216, composed by Mozart. The track will be played through two speakers on opposite sides, 30 cm away from the baby's ears, to optimize sound perception. High quality digital audio will be used to make babies listen. Music will be played at a level that can be heard in high noise pollution (i.e. the noise of incubator operation and the white noise of the recorder), but taking into account the permissible sound level recommended by the American Academy of Pediatrics, i.e. 65-70 dB
  Arms: experiment group

SUMMARY:
Bacterial meningitis is a serious infection that is more common in newborns is associated with significant morbidity and mortality. The gold standard for the diagnosis of bacterial meningitis is a positive cerebrospinal fluid (CSF) culture, usually obtained via lumbar puncture (LP). İnfants and children have similar physiological responses to pain as adults has led to greater emphasis on the assessment and management of pain in children. Therefore, management of painful interventions is important. Music may improve oxygen saturation in preterm infants undergoing endotracheal suctioning and may also reduce stress and pain in children undergoing painful medical procedures such as intravenous injections, lumbar punctures, and dental procedures. Although there are studies in the literature examining the effect of music therapy on heel blood collection or intravenous injection, no study has been found examining the effect of music therapy on the baby's pain perception during lumbar puncture. The aim of this study is to examine whether music therapy applied during lumbar puncture affects the baby's reactions to pain.

DETAILED DESCRIPTION:
Bacterial meningitis is a serious infection that is more common in newborns than in other age groups and is associated with significant morbidity and mortality. The gold standard for the diagnosis of bacterial meningitis is a positive cerebrospinal fluid (CSF) culture, usually obtained via lumbar puncture (LP). Clinical suspicion of meningitis is greater in the presence of seizures, fever, swollen fontanelle, and abnormal consciousness, but initial symptoms are often vague in the neonatal period, especially in young infants. The United States and United Kingdom guidelines recommend performing LP in newborns and infants in cases of suspected sepsis and meningitis. There have been significant changes in our understanding of the pathophysiology of pain in children over the last 20 years. There is increasing evidence to suggest that neonates as young as 24 to 25 weeks of gestation have fully developed neural pathways for the transmission and perception of pain. Additionally, exposure to pain early in life can have both immediate and long-term detrimental effects on children. The realization that infants and children have similar physiological responses to pain as adults has led to greater emphasis on the assessment and management of pain in children. Therefore, management of painful interventions is important. Various studies have proven that listening to music, sounds and heartbeats can positively affect the physiological indicators, nutrition, length of stay and pain outcomes of newborn babies. Listening to music and parents' preferred lullabies can be used to objectively determine the effects of these interventions on premature newborns' heart rate, oxygen saturation, nutrient absorption, and calorie intake. Music may improve oxygen saturation in preterm infants undergoing endotracheal suctioning and may also reduce stress and pain in children undergoing painful medical procedures such as intravenous injections, lumbar punctures, and dental procedures. Although there are studies in the literature examining the effect of music therapy on heel blood collection or intravenous injection, no study has been found examining the effect of music therapy on the baby's pain perception during lumbar puncture. The aim of this study is to examine whether music therapy applied during lumbar puncture affects the baby's reactions to pain.

ELIGIBILITY:
Inclusion Criteria:

* Having normal brainstem auditory responses
* Gestational age between 32-40
* Feeding the baby before the procedure
* Implementation of LP initiative

Exclusion Criteria:

* Having a genetic diagnosis
* Having a neurometabolic diagnosis
* Congenital malformations, mechanical ventilation, asphyxia, anomalies associated with neurological disorders, use of sedatives, or other comorbid conditions that may affect the response to musical stimuli or data collection

Ages: 32 Days to 40 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 25 (Estimated)
Dates: Start 2024-05-15 (Actual); Primary Completion 2025-11-01 (Estimated); Study Completion 2025-11-01 (Estimated)

PRIMARY OUTCOMES:
pain reduction | 40 minute
  pain relief Neonatal Infant Pain Scale (NIPS), which is a behavioral assessment tool for measuring pain in preterm and term newborns, was developed by Lawrence et al. (1993). Cronbach's alpha value was found to be 0.95 before the procedure, 0.87 during the procedure, and 0.88 after the procedure (Lawrence et al., 1993). Turkish validity and reliability were determined by Akdovan (1999). This scale was created to measure the response of the term or preterm newborn to procedural pain or distress.Parameters include babies' facial expressions, crying, breathing patterns, arm movements, leg movements, and arousal state.The total score varies between 0 and 7. Higher scores indicate higher pain levels. In other words, as the score increases, the severity of pain also increases. 0-2 points indicate no pain/mild pain, 3-4 points indicate mild pain/moderate pain, and >4 points indicate severe pain.
vital signs: O2 Saturation | 40 minute
  O2 Saturation Using an oximeter, arterial oxygen saturation (SaO2) will be measured and recorded from 10 minutes before the procedure until the end of the procedure. Babies' oxygen saturations will be measured with a pulse oximeter placed on the wrist and monitored. All babies in the neonatal intensive care unit are constantly monitored with a monitor device. The will be monitored and recorded using this monitor. The value will be recorded 10 minutes before the transaction, during the transaction, 10 minutes after the transaction and 20 minutes after the transaction.
vital signs: Heart rate | 40 minute
  Heart rate (beats per minute) All babies in the neonatal intensive care unit are constantly monitored with a monitor device. The babies' heart rate per minute will be monitored and recorded using this monitor. The value will be recorded 10 minutes before the transaction, during the transaction, 10 minutes after the transaction and 20 minutes after the transaction.
baby's crying duration (sec) | 40 minute
  During the procedure, the baby's crying time will be tracked and recorded in seconds.

CONTACTS AND LOCATIONS:
Overall Officials: Ayşe Metin, phd, Study Chair — kutuphane@erzurum.edu.tr
Locations (1):
- Ayşe Metin, Erzurum, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No